CLINICAL TRIAL: NCT03789149
Title: Focal Intraoperative Radiotherapy After Resection of Brain Metastases
Brief Title: Focal Intraoperative Radiotherapy of Brain Metastases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Planning to join a prospective multicentric trial after evaluation of 10 first participants
Sponsor: AC Camargo Cancer Center (Other)
Collaborators: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2315/17
Record Dates: First submitted 2018-12-26; First posted 2018-12-28 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-07

CONDITIONS: Brain Metastases, Adult; Central Nervous System Metastases
Keywords: Intraoperative Radiotherapy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intraoperative Radiotherapy (Experimental): Intraoperative Radiotherapy with a mobile device (Intrabeam, Carl Zeiss AG)
  Interventions: Radiation: Intraoperative Radiotherapy

INTERVENTIONS:
Radiation: Intraoperative Radiotherapy — Intraoperative Radiotherapy with a mobile device (Intrabeam, Carl Zeiss AG) consisting of a small source of low energy x-rays (30-50 kV) mounted on a mechanical arm with six degrees of freedom. The resulting dose distribution is isotropic around the tip of the X-ray source. A set of spherical applicators with diameters ranging from 1.5 to 5 cm is available to connect to the source. The treatment time may vary from 20-30 minutes with the suggested dose of 18 Gy to the resection cavity to a depth of 1 mm.
  Other Names: Intrabeam

SUMMARY:
Brain metastases (BM) are the most prevalent tumors of the central nervous system (CNS), with a ratio of 10: 1 in relation to primary tumors. In prospective studies, whole-brain radiotherapy (WBRT) reduced the risk of local recurrence after resection of brain metastases from 46-59% to 10-28%. Furthermore, WBRT reduces the incidence of new metastases and death from disease, but no apparent improvement in overall survival (OS). Due to the potential neurocognitive effects associated with WBRT compared to isolated focal approach, several authors have suggested delaying WBRT and perform focal adjuvant RT after resection of isolated BM. In this context, intraoperative radiotherapy (IORT) in the cavity after resection of BM may be an appealing option.

The primary objectives of this study are to evaluate local control (LC) and the control of brain disease (LC associated with the absence of new distant BM) after IORT for one completely resected supratentorial BM in the presence of up to 10 lesions suggestive of BM.

DETAILED DESCRIPTION:
Brain metastases (BM) are the most prevalent tumors of the central nervous system (CNS), with a ratio of 10: 1 in relation to primary tumors. This type of metastasis occurs in 20-40% of cancer patients and are related to significant morbidity and mortality.

In prospective studies, whole-brain radiotherapy (WBRT) reduced the risk of local recurrence after resection of brain metastases from 46-59% to 10-28%. Furthermore, WBRT reduces the incidence of new metastases and death from disease, but no apparent improvement in overall survival (OS). Due to the potential neurocognitive effects associated with WBRT compared to isolated focal approach, several authors have suggested delaying WBRT and perform focal adjuvant RT after resection of isolated BM.

The utilization of intraoperative radiotherapy (IORT) in the cavity after resection of primary or BM has been described in the literature, the majority of reports describes performing brachytherapy with iodine seeds or interstitial radiosurgery. However, there is a paucity of information regarding the use of IORT with low energy X-ray for focal treatment after resection of brain BM.

The objectives of this study are evaluate local control (LC), the control of brain disease in patients with metastatic brain disease (up to 10 lesions) submitted to focal IORT to an isolated surgical cavity, evaluate overall survival (OS), evaluate the frequency of radiation necrosis and correlate the prognostic factors related to the patient with OS and the parameters of the treatment (dose, volume, lesion location) with the LC and radiation necrosis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Histologically confirmed diagnosis of invasive cancer in the presence of up to 10 lesions suggestive of BM
* Indication of resection of single lesion suggestive of BM and evidence of macroscopic complete resection
* Patient consent to participate in the study

Exclusion Criteria:

* Previous cranial radiotherapy
* Any kind of antineoplasic systemic treatment for less than 7 days of the procedure
* Cavities with proximity < 10 mm from the brainstem or optical pathway.
* Pregnant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Local control (LC) | 1 year
  Rate of local failure in the surgical cavity
Control of Brain Disease (CBD) | 1 year
  Rate of control in the brain outside

SECONDARY OUTCOMES:
Overall Survival (OS) | 1 year
  Rate of death related to any cause
Frequency of radiation necrosis | 1 year
  Imaging evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Douglas G Castro, MD, Principal Investigator — AC Camargo Cancer Center
Locations (1):
- AC Camargo Cancer Center, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR
Time Frame: 6 months after publication
Access Criteria: Correlated Area Investigators with publishing background and a defined objective